CLINICAL TRIAL: NCT02504216
Title: An International, Multicenter, Randomized, Double-blind, Placebo-controlled Phase 3 Trial Investigating the Efficacy and Safety of Rivaroxaban to Reduce the Risk of Major Thrombotic Vascular Events in Patients With Symptomatic Peripheral Artery Disease Undergoing Lower Extremity Revascularization Procedures
Brief Title: Efficacy and Safety of Rivaroxaban in Reducing the Risk of Major Thrombotic Vascular Events in Subjects With Symptomatic Peripheral Artery Disease Undergoing Peripheral Revascularization Procedures of the Lower Extremities
Acronym: VOYAGER PAD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Janssen Research & Development, LLC (Industry); Colorado Prevention Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 17454; 2014-005569-58 (EudraCT Number)
Record Dates: First submitted 2015-07-20; First posted 2015-07-21 (Estimated); Results first posted 2020-12-08 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Peripheral Artery Disease
Keywords: Rivaroxaban; Xarelto; Aspirin; Acetylic salicylic acid; Anticoagulant; Peripheral artery disease; Peripheral arterial disease; Revascularization; Acute limb ischemia; Amputation; Cardiovascular events
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Rivaroxaban

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Rivaroxaban (Experimental): Rivaroxaban 2.5 mg orally twice daily (5 mg cumulative daily dose)
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939)
- Placebo (Placebo Comparator): Rivaroxaban-placebo orally twice daily
  Interventions: Drug: Rivaroxaban-Placebo

INTERVENTIONS:
Drug: Rivaroxaban (Xarelto, BAY59-7939) — 2.5 mg, twice daily, orally, tablet
  Arms: Rivaroxaban
Drug: Rivaroxaban-Placebo — matching placebo, twice daily, orally, tablet
  Arms: Placebo

SUMMARY:
The purpose of study was to test whether rivaroxaban added to standard of care treatment, when compared to placebo, had the potential to reduce the incidence of the clinical events related to the clots and complications of the heart and brain (CV death, MI, or stroke) or the legs (acute limb ischemia or major amputation) in patients who had undergone recent procedure(s) to improve the blood flow of their legs.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥50
* Documented moderate to severe symptomatic lower extremity atherosclerotic peripheral artery disease
* Technically successful peripheral revascularization distal to the external iliac artery for symptomatic PAD (Peripheral artery disease) within the last 10 days prior to randomization

Exclusion Criteria:

* Patients undergoing revascularization for asymptomatic PAD or mild claudication without functional limitation of the index leg.
* Patients undergoing revascularization of the index leg to treat an asymptomatic or minimally symptomatic restenosis of a bypass graft or target lesion restenosis.
* Prior revascularization on the index leg within 10 days of the qualifying revascularization.
* Planned dual antiplatelet therapy (DAPT) use for the qualifying revascularization procedure of clopidogrel in addition to Acetylic salicylic acid (ASA) for >6 months after the qualifying revascularization procedure; it is strongly recommended that any course of clopidogrel is kept to the minimum necessary in accordance with local standard of care and international practice guidelines (typically 30 days, or up to 60 days for some drug-coated products or devices) and is only allowed for up to 6 months for complex procedures or devices in the investigator's opinion that require longer use.
* Planned use of any additional antiplatelet agent other than clopidogrel and ASA after the qualifying revascularization procedure.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6564 (Actual)
Dates: Start 2015-08-18 (Actual); Primary Completion 2019-11-27 (Actual); Study Completion 2020-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (426):
- United States (94):
  - Alexander City, Alabama
  - Birmingham, Alabama
  - Fort Payne, Alabama
  - Huntsville, Alabama
  - Avondale, Arizona
  - Glendale, Arizona
  - Phoenix, Arizona
  - Mission Viejo, California
  - Northridge, California
  - Palo Alto, California
  - Roseville, California
  - Stanford, California
  - Torrance, California
  - Aurora, Colorado
  - Denver, Colorado
  - Washington D.C., District of Columbia
  - Atlantis, Florida
  - Clearwater, Florida
  - Daytona Beach, Florida
  - Gainesville, Florida
  - Hudson, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Ocala, Florida
  - Pensacola, Florida
  - Safety Harbor, Florida
  - Tallahassee, Florida
  - Wellington, Florida
  - Arlington Heights, Illinois
  - Elk Grove Village, Illinois
  - Springfield, Illinois
  - Urbana, Illinois
  - Fort Wayne, Indiana
  - Merrillville, Indiana
  - Iowa City, Iowa
  - Lexington, Kentucky
  - Alexandria, Louisiana
  - Covington, Louisiana
  - Shreveport, Louisiana
  - Lewiston, Maine
  - Baltimore, Maryland
  - Clinton, Maryland
  - Bay City, Michigan
  - Dearborn, Michigan
  - Detroit, Michigan
  - Lansing, Michigan
  - Midland, Michigan
  - Muskegon, Michigan
  - Wyoming, Michigan
  - Coon Rapids, Minnesota
  - Saint Cloud, Minnesota
  - Jackson, Mississippi
  - Tupelo, Mississippi
  - Springfield, Missouri
  - St Louis, Missouri
  - Lincoln, Nebraska
  - Lebanon, New Hampshire
  - Flemington, New Jersey
  - Linden, New Jersey
  - Teaneck, New Jersey
  - New York, New York
  - Saratoga Springs, New York
  - Chapel Hill, North Carolina
  - Charlotte, North Carolina
  - Durham, North Carolina
  - Winston-Salem, North Carolina
  - Minot, North Dakota
  - Cincinnati, Ohio
  - Dayton, Ohio
  - Springfield, Ohio
  - Toledo, Ohio
  - Oklahoma City, Oklahoma
  - Hillsboro, Oregon
  - Camp Hill, Pennsylvania
  - Erie, Pennsylvania
  - Philadelphia, Pennsylvania
  - York, Pennsylvania
  - Greenville, South Carolina
  - Rapid City, South Dakota
  - Knoxville, Tennessee
  - Amarillo, Texas
  - Austin, Texas
  - Dallas, Texas
  - Edinburg, Texas
  - Houston, Texas
  - Humble, Texas
  - Huntsville, Texas
  - Kingwood, Texas
  - San Antonio, Texas
  - Tyler, Texas
  - Victoria, Texas
  - Madison, Wisconsin
  - Manitowoc, Wisconsin
  - Wausau, Wisconsin
- Argentina (15):
  - Bahía Blanca, Buenos Aires
  - Ciudadela, Buenos Aires
  - Coronel Suárez, Buenos Aires
  - Junín, Buenos Aires
  - La Plata, Buenos Aires
  - Mar del Plata, Buenos Aires
  - San Isidro, Buenos Aires
  - San Martín, Buenos Aires
  - Buenos Aires, Ciudad Auton. de Buenos Aires
  - Santa Rosa, La Pampa Province
  - Rosario, Santa Fe Province
  - Ciudad Auton. de Buenos Aires
  - Corrientes
  - Córdoba
  - Santa Fe
- Austria (6):
  - Klagenfurt, Carinthia
  - Graz, Styria
  - Innsbruck, Tyrol
  - Feldkirch, Vorarlberg
  - Linz
  - Vienna
- Belgium (5):
  - Bruxelles - Brussel
  - Genk
  - Ghent
  - Kortrijk
  - Leuven
- Brazil (15):
  - Fortaleza, Ceará
  - Belo Horizonte, Minas Gerais
  - Uberlândia, Minas Gerais
  - Curitiba, Paraná
  - Canoas, Rio Grande do Sul
  - Passo Fundo, Rio Grande do Sul
  - Porto Alegre, Rio Grande do Sul
  - Belo Horizonte, São Paulo
  - Campinas, São Paulo
  - Santo André, São Paulo
  - São Bernardo do Campo, São Paulo
  - São José do Rio Preto, São Paulo
  - São Paulo, São Paulo
  - Tatuí, São Paulo
  - Rio de Janeiro
- Bulgaria (9):
  - Burgas
  - Panagyurishte
  - Plovdiv
  - Rousse
  - Samokov
  - Sofia
  - Stara Zagora
  - Varna
  - Yambol
- Canada (11):
  - Winnipeg, Manitoba
  - St. John's, Newfoundland and Labrador
  - Hamilton, Ontario
  - London, Ontario
  - Ottawa, Ontario
  - Chicoutimi, Quebec
  - Gatineau, Quebec
  - Montreal, Quebec
  - Saint-Jérôme, Quebec
  - Québec
  - Vancouver
- China (21):
  - Hefei, Anhui
  - Chongqing, Chongqing Municipality
  - Fuzhou, Fujian
  - Zhangzhou, Fujian
  - Guangzhou, Guangdong
  - Zhanjiang, Guangdong
  - Zhongshan, Guangdong
  - Haikou, Hainan
  - Wuhan, Hubei
  - Changsha, Hunan
  - Changzhou, Jiangsu
  - Nanjing, Jiangsu
  - Changchun, Jilin
  - Xi'an, Shaanxi
  - Qingdao, Shandong
  - Taiyuan, Shanxi
  - Taizhou, Zhejiang
  - Wenzhou, Zhejiang
  - Beijing
  - Shanghai
  - Tianjin
- Czechia (10):
  - Brno
  - Hodonín
  - Hradec Králové
  - Kladno
  - Liberec
  - Olomouc
  - Pilsen
  - Prague
  - Prostějov
  - Vratimov
- Denmark (5):
  - Aarhus N
  - Kolding
  - København Ø
  - Odense C
  - Viborg
- Estonia (2):
  - Tallinn
  - Tartu
- Finland (3):
  - Helsinki
  - Oulu
  - Tampere
- France (13):
  - Bordeaux
  - Caen
  - Castelnau-le-Lez
  - Grenoble
  - Le Coudray
  - Limoges
  - Montpellier
  - Nice
  - Paris
  - Poitiers
  - Rennes
  - Strasbourg
  - Toulouse
- Germany (34):
  - Bad Friedrichshall, Baden-Wurttemberg
  - Bad Krozingen, Baden-Wurttemberg
  - Freudenstadt, Baden-Wurttemberg
  - Heidelberg, Baden-Wurttemberg
  - Karlsbad, Baden-Wurttemberg
  - Karlsruhe, Baden-Wurttemberg
  - Ulm, Baden-Wurttemberg
  - Erlangen, Bavaria
  - Immenstadt im Allgäu, Bavaria
  - München, Bavaria
  - Regensburg, Bavaria
  - Rosenheim, Bavaria
  - Bad Nauheim, Hesse
  - Darmstadt, Hesse
  - Frankfurt am Main, Hesse
  - Arnsberg, North Rhine-Westphalia
  - Bielefeld, North Rhine-Westphalia
  - Cologne, North Rhine-Westphalia
  - Düsseldorf, North Rhine-Westphalia
  - Krefeld, North Rhine-Westphalia
  - Münster, North Rhine-Westphalia
  - Wesel, North Rhine-Westphalia
  - Kaiserslautern, Rhineland-Palatinate
  - Mainz, Rhineland-Palatinate
  - Dresden, Saxony
  - Leipzig, Saxony
  - Magdeburg, Saxony-Anhalt
  - Lübeck, Schleswig-Holstein
  - Jena, Thuringia
  - Sonneberg, Thuringia
  - Berlin
  - Bremen
  - Dresden
  - Hamburg
- Hungary (11):
  - Budapest
  - Debrecen
  - Győr
  - Kaposvár
  - Kistarcsa
  - Miskolc
  - Nyíregyháza
  - Pécs
  - Szeged
  - Székesfehérvár
  - Szombathely
- Italy (16):
  - Lecce, Apulia
  - Potenza, Basilicate
  - Avellino, Campania
  - Napoli, Campania
  - Bologna, Emilia-Romagna
  - Ravenna, Emilia-Romagna
  - Reggio Emilia, Emilia-Romagna
  - Rome, Lazio
  - Milan, Lombardy
  - Varese, Lombardy
  - Turin, Piedmont
  - Palermo, Sicily
  - Ragusa, Sicily
  - Macerata, The Marches
  - Florence, Tuscany
  - Perugia, Umbria
- Japan (40):
  - Nagakute, Aichi-ken
  - Matsuyama, Ehime
  - Kitakyushu, Fukuoka
  - Kurume, Fukuoka
  - Shibukawa, Gunma
  - Hatsukaichi, Hiroshima
  - Asahikwa, Hokkaido
  - Sapporo, Hokkaido
  - Tomakomai, Hokkaido
  - Amagasaki, Hyōgo
  - Himeji, Hyōgo
  - Kobe, Hyōgo
  - Takarazuka, Hyōgo
  - Morioka, Iwate
  - Takamatsu, Kagawa-ken
  - Kawasaki, Kanagawa
  - Sagamihara, Kanagawa
  - Matsusaka, Mie-ken
  - Matsumoto, Nagano
  - Kashihara, Nara
  - Beppu, Oita Prefecture
  - Habikino, Osaka
  - Kawagoe, Saitama
  - Ōmihachiman, Shiga
  - Hamada, Shimane
  - Bunkyo-ku, Tokyo
  - Fuchū, Tokyo
  - Itabashi-ku, Tokyo
  - Meguro-ku, Tokyo
  - Minato, Tokyo
  - Minato-ku, Tokyo
  - Suginami-ku, Tokyo
  - Gifu
  - Kagoshima
  - Kumamoto
  - Kyoto
  - Miyazaki
  - Osaka
  - Saitama
  - Shizuoka
- Latvia (3):
  - Daugavpils
  - Liepāja
  - Riga
- Lithuania (3):
  - Kaunas
  - Panevezys
  - Vilnius
- Netherlands (7):
  - 's-Hertogenbosch
  - Eindhoven
  - Enschede
  - Heerlen
  - Utrecht
  - Veldhoven
  - Zwolle
- Poland (11):
  - Bialystok
  - Bydgoszcz
  - Gdynia
  - Katowice
  - Krakow
  - Lodz
  - Lublin
  - Poznan
  - Szczecin
  - Warsaw
  - Wroclaw
- Portugal (5):
  - Almada, Setúbal District
  - Lisbon
  - Ponta Delgada
  - Porto
  - Vila Nova de Gaia
- Romania (7):
  - Piteşti, Argeş
  - Bucharest
  - Cluj-Napoca
  - Iași
  - Oradea
  - Târgu Mureş
  - Timișoara
- Russia (10):
  - Kemerovo
  - Moscow
  - Nizhny Novgorod
  - Novosibirsk
  - Rostov-on-Don
  - Ryazan
  - Saint Petersburg
  - Tomsk
  - Tver'
  - Voronezh
- Serbia (2):
  - Belgrade
  - Niš
- Slovakia (8):
  - Bardejov
  - Bratislava
  - Dunajská Streda
  - Košice
  - Nitra
  - Nové Zámky
  - Trnava
  - Žilina
- South Korea (8):
  - Goyang-si, Gyeonggido
  - Seongnam-si, Gyeonggido
  - Incheon, Incheon Gwang''yeogsi
  - Busan
  - Daegu
  - Daejeon
  - Jung-gu Daejeon
  - Seoul
- Spain (10):
  - Cadiz, Andalusia
  - L'Hospitalet de Llobregat, Barcelona
  - Sabadell, Barcelona
  - A Coruña
  - Barcelona
  - Ciudad Real
  - Granada
  - Madrid
  - Pamplona
  - Tarragona
- Sweden (5):
  - Gothenburg
  - Linköping
  - Malmo
  - Solna
  - Vaxjo
- Switzerland (8):
  - Basel, Canton of Basel-City
  - Sankt Gallen, Canton of St. Gallen
  - Chur, Kanton Graubünden
  - Baden
  - Bern
  - Fribourg
  - Geneva
  - Lucerne
- Taiwan (5):
  - Hsinchu
  - Kaohsiung City
  - Tainan
  - Taipei
  - Taoyuan District
- Thailand (3):
  - Bangkok
  - Khon Kaen
  - Songkhla
- Ukraine (8):
  - Dnipro
  - Ivano-Frankivsk
  - Kharkiv
  - Kiev
  - Kyiv
  - Lviv
  - Vinnytsia
  - Zaporizhzhya
- United Kingdom (13):
  - Carlisle, Cumbria
  - Hull, Humberside
  - Harrow, London
  - Doncaster, South Yorkshire
  - Newcastle upon Tyne, Tyne and Wear
  - Birmingham, West Midlands
  - Leeds, West Yorkshire
  - Worcester, Worcestershire
  - Cambridge
  - Cheltenham
  - London
  - Manchester
  - Sheffield

REFERENCES:
- [Derived] Hogan S, Szarek M, Debus ES, Nehler M, Anand SS, Patel MR, Pap AF, Deng H, Hodge S, Haskell LP, Muehlhofer E, Berkowitz SE, Bauersachs RM, Bonaca MP. Rivaroxaban in Peripheral Artery Disease After Revascularization: Worst Events and Net Outcomes in VOYAGER PAD. J Am Heart Assoc. 2025 Nov 4;14(21):e039752. doi: 10.1161/JAHA.124.039752. Epub 2025 Oct 23. PMID 41128134
- [Derived] Rogers RK, Herold J, Govsyeyev N, Iezzi R, Morrison J, Hogan SE, Nehler M, Bricker R, Andring B, Bergmark B, Cavender M, Malgor E, Jacobs D, Young MN, Capell W, Ycas JW, Anand SS, Berkowitz SD, Debus ES, Haskell LP, Muehlhofer E, Patel MR, Hess CN, Bauersachs RM, Anderson V, Bonaca MP. Methods, design, and initial results of an angiographic core lab from VOYAGER-PAD. Vasc Med. 2024 Apr;29(2):143-152. doi: 10.1177/1358863X241228542. Epub 2024 Mar 17. PMID 38493348
- [Derived] Hogan SE, Debus ES, Nehler MR, Patel MR, Anand SS, Muehlhofer E, Haskell LP, Berkowitz SD, Bauersachs RM, Bonaca MP. Unplanned Index Limb Revascularization With Rivaroxaban Versus Placebo in Patients With Critical Limb-Threatening Ischemia After Endovascular and Surgical Treatment: Insights From VOYAGER PAD. Circulation. 2024 Feb 20;149(8):635-637. doi: 10.1161/CIRCULATIONAHA.123.065330. Epub 2024 Feb 20. No abstract available. PMID 38377256
- [Derived] Govsyeyev N, Nehler M, Conte MS, Debus S, Chung J, Dorigo W, Gudz I, Krievins D, Mills J, Moll F, Norgren L, Piffaretti G, Powell R, Szalay D, Sillesen H, Wohlauer M, Szarek M, Bauersachs RM, Anand SS, Patel MR, Capell WH, Jaeger N, Hess CN, Muehlhofer E, Haskell LP, Berkowitz SD, Bonaca MP. Rivaroxaban in patients with symptomatic peripheral artery disease after lower extremity bypass surgery with venous and prosthetic conduits. J Vasc Surg. 2023 Apr;77(4):1107-1118.e2. doi: 10.1016/j.jvs.2022.11.062. Epub 2022 Dec 5. PMID 36470531
- [Derived] Hess CN, Baumgartner I, Anand SS, Nehler MR, Patel MR, Debus ES, Szarek M, Capell W, Muehlhofer E, Berkowitz SD, Haskell LP, Bauersachs RM, Bonaca MP, Hsia J. Sex-Based Differences in Outcomes Following Peripheral Artery Revascularization: Insights From VOYAGER PAD. J Am Heart Assoc. 2022 Jun 21;11(12):e024655. doi: 10.1161/JAHA.121.024655. Epub 2022 Jun 14. PMID 35699170
- [Derived] Hogan SE, Nehler MR, Anand S, Patel MR, Debus S, Jackson MT, Buchanan C, King RW, Hess C, Muehlhofer E, Haskell LP, Bauersachs RM, Berkowitz SD, Hsia J, Bonaca MP. Improvement in walking impairment following surgical and endovascular revascularization: Insights from VOYAGER PAD. Vasc Med. 2022 Aug;27(4):343-349. doi: 10.1177/1358863X221085606. Epub 2022 Apr 25. PMID 35467452
- [Derived] Hess CN, Patel MR, Bauersachs RM, Anand SS, Debus ES, Nehler MR, Fanelli F, Yeh RW, Secemsky EA, Beckman JA, Mauri L, Govsyeyev N, Capell WH, Brackin T, Berkowitz SD, Muehlhofer E, Haskell LP, Hiatt WR, Bonaca MP. Safety and Effectiveness of Paclitaxel Drug-Coated Devices in Peripheral Artery Revascularization: Insights From VOYAGER PAD. J Am Coll Cardiol. 2021 Nov 2;78(18):1768-1778. doi: 10.1016/j.jacc.2021.08.052. PMID 34711335
- [Derived] Debus ES, Nehler MR, Govsyeyev N, Bauersachs RM, Anand SS, Patel MR, Fanelli F, Capell WH, Brackin T, Hinterreiter F, Krievins D, Nault P, Piffaretti G, Svetlikov A, Jaeger N, Hess CN, Sillesen HH, Conte M, Mills J, Muehlhofer E, Haskell LP, Berkowitz SD, Hiatt WR, Bonaca MP. Effect of Rivaroxaban and Aspirin in Patients With Peripheral Artery Disease Undergoing Surgical Revascularization: Insights From the VOYAGER PAD Trial. Circulation. 2021 Oct 5;144(14):1104-1116. doi: 10.1161/CIRCULATIONAHA.121.054835. Epub 2021 Aug 12. PMID 34380322
- [Derived] Bauersachs RM, Szarek M, Brodmann M, Gudz I, Debus ES, Nehler MR, Anand SS, Patel MR, Hess CN, Capell WH, Rogers K, Muehlhofer E, Haskell LP, Berkowitz SD, Hiatt WR, Bonaca MP; VOYAGER PAD Committees and Investigators. Total Ischemic Event Reduction With Rivaroxaban After Peripheral Arterial Revascularization in the VOYAGER PAD Trial. J Am Coll Cardiol. 2021 Jul 27;78(4):317-326. doi: 10.1016/j.jacc.2021.05.003. Epub 2021 May 16. PMID 34010631
- [Derived] Hiatt WR, Bonaca MP, Patel MR, Nehler MR, Debus ES, Anand SS, Capell WH, Brackin T, Jaeger N, Hess CN, Pap AF, Berkowitz SD, Muehlhofer E, Haskell L, Brasil D, Madaric J, Sillesen H, Szalay D, Bauersachs R. Rivaroxaban and Aspirin in Peripheral Artery Disease Lower Extremity Revascularization: Impact of Concomitant Clopidogrel on Efficacy and Safety. Circulation. 2020 Dec 8;142(23):2219-2230. doi: 10.1161/CIRCULATIONAHA.120.050465. Epub 2020 Nov 3. PMID 33138628
- [Derived] Bonaca MP, Bauersachs RM, Anand SS, Debus ES, Nehler MR, Patel MR, Fanelli F, Capell WH, Diao L, Jaeger N, Hess CN, Pap AF, Kittelson JM, Gudz I, Matyas L, Krievins DK, Diaz R, Brodmann M, Muehlhofer E, Haskell LP, Berkowitz SD, Hiatt WR. Rivaroxaban in Peripheral Artery Disease after Revascularization. N Engl J Med. 2020 May 21;382(21):1994-2004. doi: 10.1056/NEJMoa2000052. Epub 2020 Mar 28. PMID 32222135
- [Derived] Capell WH, Bonaca MP, Nehler MR, Chen E, Kittelson JM, Anand SS, Berkowitz SD, Debus ES, Fanelli F, Haskell L, Patel MR, Bauersachs R, Hiatt WR. Rationale and design for the Vascular Outcomes study of ASA along with rivaroxaban in endovascular or surgical limb revascularization for peripheral artery disease (VOYAGER PAD). Am Heart J. 2018 May;199:83-91. doi: 10.1016/j.ahj.2018.01.011. Epub 2018 Feb 3. PMID 29754671

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at 548 centers which screened participants (534 sites randomized participants) worldwide between 18 Aug 2015 (first patient's first visit) and 27 Nov 2019 (last patient's last visit).
Pre-assignment Details: A total of 6772 participants were screened, of which 6564 were randomly assigned to either of the two treatment arms.
Groups:
- Rivaroxaban 2.5 mg Bid + Aspirin 100 mg od: Participants were treated with Rivaroxaban 2.5 mg twice-daily (bid) and aspirin (ASA: Acetylsalicylic Acid) 100 mg once-daily (od)
- Rivaroxaban Placebo Bid + Aspirin 100 mg od: Participants were treated with Rivaroxaban-placebo twice-daily and aspirin (ASA: Acetylsalicylic Acid) 100 mg once-daily
Period: Overall Study
Arm/Group | Rivaroxaban 2.5 mg Bid + Aspirin 100 mg od | Rivaroxaban Placebo Bid + Aspirin 100 mg od
Started | 3286 | 3278
Received Treatment | 3256 | 3248
Completed (Vital status known at ECOD) | 3275 | 3263
Not Completed | 11 | 15
Not completed — Lost to Follow-up | 3 | 3
Not completed — Withdrawal by Subject | 8 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rivaroxaban 2.5 mg Bid + Aspirin 100 mg od | Rivaroxaban Placebo Bid + Aspirin 100 mg od | Total
Number analyzed (Participants) | 3286 | 3278 | 6564
Age, Continuous [Median (Full Range); unit: Years] | 67.0 [49 to 93] | 67.0 [50 to 95] | 67 [49 to 95]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 847 | 857 | 1704
  Male | 2439 | 2421 | 4860
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 4 | 5
  Asian | 484 | 482 | 966
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 84 | 71 | 155
  White | 2647 | 2656 | 5303
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 69 | 62 | 131

OUTCOME MEASURES:

1. Primary Outcome: Primary Efficacy Outcome: Number of Participants With Composite of Myocardial Infarction (MI), Ischemic Stroke, Cardiovascular Death, Acute Limb Ischemia (ALI) and Major Amputation Due to a Vascular Etiology
Description: Only the first occurrence of the outcome event under analysis within the data scope from a participant is considered.
Time Frame: For each participant, the first occurrence of the composite primary efficacy outcome after randomization up until the efficacy cut-off date (08-Sep-2019) was considered. The mean time in follow-up survival time until ECOD that date was 1109.76 days.
Population: Intention-to-treat analysis set (ITT Set): Comprised all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Rivaroxaban 2.5 mg Bid + Aspirin 100 mg od | Rivaroxaban Placebo Bid + Aspirin 100 mg od
Number analyzed (Participants) | 3286 | 3278
Participants | 508 | 584
Statistical Analysis 1: Comparison: Rivaroxaban 2.5 mg Bid + Aspirin 100 mg od vs Rivaroxaban Placebo Bid + Aspirin 100 mg od; IxRS: Interactive web/voice response system; Test type: Superiority; p = 0.0043, Log Rank; P-value (1-sided) is based on the log rank test stratified by type of procedure and clopidogrel use per IxRS assignment with treatment as a factor; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.76 to 0.96]

2. Primary Outcome: Primary Safety Outcome: Number of Participants With TIMI (Thrombolysis in Myocardial Infarction) Major Bleeding
Description: Only the first occurrence of the outcome event under analysis within the data scope from a participant is considered.
Time Frame: For each participant, the first occurrence of the primary safety outcome after randomization up until 2 days after permanent stop of study drug (rivaroxaban or rivaroxaban placebo).
Population: Safety analysis set (SAF Set): Comprised all treated participants, i.e. randomized participants who received at least one dose of study drug (rivaroxaban or rivaroxaban placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Rivaroxaban 2.5 mg Bid + Aspirin 100 mg od | Rivaroxaban Placebo Bid + Aspirin 100 mg od
Number analyzed (Participants) | 3256 | 3248
Participants | 62 | 44
Statistical Analysis 1: Comparison: Rivaroxaban 2.5 mg Bid + Aspirin 100 mg od vs Rivaroxaban Placebo Bid + Aspirin 100 mg od; Test type: Other; p = 0.0695, Log Rank; P-value (2-sided) is based on the log rank test stratified by type of procedure and clopidogrel use per IxRS assignment with treatment as a factor; Hazard Ratio (HR) = 1.43, 95% CI 2-sided [0.97 to 2.10]

3. Secondary Outcome: Number of Participants With Composite of MI, Ischemic Stroke, Coronary Heart Disease (CHD) Death, ALI, and Major Amputation of a Vascular Etiology
Description: Only the first occurrence of the outcome event under analysis within the data scope from a participant is considered.
Time Frame: For each participant, the first occurrence of the composite efficacy outcome after randomization up until the efficacy cut-off date (08-Sep-2019) was considered. The mean survival time until ECOD was 1108.79 days.
Population: Intention-to-treat analysis set (ITT Set): Comprised all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Rivaroxaban 2.5 mg Bid + Aspirin 100 mg od | Rivaroxaban Placebo Bid + Aspirin 100 mg od
Number analyzed (Participants) | 3286 | 3278
Participants | 433 | 528
Statistical Analysis 1: Comparison: Rivaroxaban 2.5 mg Bid + Aspirin 100 mg od vs Rivaroxaban Placebo Bid + Aspirin 100 mg od; Test type: Superiority; p = 0.0004, Log Rank — P-value (1-sided) is based on the log rank test stratified by type of procedure and clopidogrel use per IxRS assignment with treatment as a factor; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.71 to 0.91]

4. Secondary Outcome: Number of Participants With an Unplanned Index Limb Revascularization for Recurrent Limb Ischemia (Subsequent Index Leg Revascularization That Was Not Planned or Considered as Part of the Initial Treatment Plan at the Time of Randomization)
Description: Only the first occurrence of the outcome event under analysis within the data scope from a participant is considered.
Time Frame: For each participant, the first occurrence of the efficacy outcome after randomization up until the efficacy cut-off date (08-Sep-2019) was considered. The mean survival time until ECOD was 1062.48 days.
Population: Intention-to-treat analysis set (ITT Set): Comprised all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Rivaroxaban 2.5 mg Bid + Aspirin 100 mg od | Rivaroxaban Placebo Bid + Aspirin 100 mg od
Number analyzed (Participants) | 3286 | 3278
Participants | 584 | 655
Statistical Analysis 1: Comparison: Rivaroxaban 2.5 mg Bid + Aspirin 100 mg od vs Rivaroxaban Placebo Bid + Aspirin 100 mg od; Test type: Superiority; p = 0.0140, Log Rank — [p-value comment as in outcome 3, analysis 1]; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.79 to 0.99]

5. Secondary Outcome: Number of Participants With Hospitalization for a Coronary or Peripheral Cause (Either Lower Limb) of a Thrombotic Nature
Description: Only the first occurrence of the outcome event under analysis within the data scope from a participant is considered.
Time Frame: For each participant, the first occurrence of the efficacy outcome after randomization up until the efficacy cut-off date (08-Sep-2019) was considered. The mean survival time until ECOD was 1154.04 days
Population: Intention-to-treat analysis set (ITT Set): Comprised all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Rivaroxaban 2.5 mg Bid + Aspirin 100 mg od | Rivaroxaban Placebo Bid + Aspirin 100 mg od
Number analyzed (Participants) | 3286 | 3278
Participants | 262 | 356
Statistical Analysis 1: Comparison: Rivaroxaban 2.5 mg Bid + Aspirin 100 mg od vs Rivaroxaban Placebo Bid + Aspirin 100 mg od; Test type: Superiority; p < 0.0001, Log Rank — [p-value comment as in outcome 3, analysis 1]; Hazard Ratio (HR) = 0.72, 95% CI 2-sided [0.62 to 0.85]

6. Secondary Outcome: Number of Participants With Composite of MI, Ischemic Stroke, All-cause Mortality (ACM), ALI, and Major Amputation of a Vascular Etiology
Description: Only the first occurrence of the outcome event under analysis within the data scope from a participant is considered.
Time Frame: For each participant, the first occurrence of the composite efficacy outcome after randomization up until the efficacy cut-off date (08-Sep-2019) was considered. The mean survival time until ECOD was 1085.13 days
Population: Intention-to-treat analysis set (ITT Set): Comprised all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Rivaroxaban 2.5 mg Bid + Aspirin 100 mg od | Rivaroxaban Placebo Bid + Aspirin 100 mg od
Number analyzed (Participants) | 3286 | 3278
Participants | 614 | 679
Statistical Analysis 1: Comparison: Rivaroxaban 2.5 mg Bid + Aspirin 100 mg od vs Rivaroxaban Placebo Bid + Aspirin 100 mg od; Test type: Superiority; p = 0.0145, Log Rank — [p-value comment as in outcome 3, analysis 1]; Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.79 to 0.99]

7. Secondary Outcome: Number of Participants With Composite of MI, All-cause Stroke, Cardiovascular (CV) Death, Acute Limb Ischemia (ALI), and Major Amputation of a Vascular Etiology
Description: Only the first occurrence of the outcome event under analysis within the data scope from a participant is considered.
Time Frame: For each participant, the first occurrence of the composite efficacy outcome after randomization up until the efficacy cut-off date (08-Sep-2019) was considered. The mean survival time until ECOD was 1108.29 days
Population: Intention-to-treat analysis set (ITT Set): Comprised all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Rivaroxaban 2.5 mg Bid + Aspirin 100 mg od | Rivaroxaban Placebo Bid + Aspirin 100 mg od
Number analyzed (Participants) | 3286 | 3278
Participants | 514 | 588
Statistical Analysis 1: Comparison: Rivaroxaban 2.5 mg Bid + Aspirin 100 mg od vs Rivaroxaban Placebo Bid + Aspirin 100 mg od; Test type: Superiority; p = 0.0051, Log Rank — [p-value comment as in outcome 3, analysis 1]; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.76 to 0.96]

8. Secondary Outcome: Number of Mortality (All-cause)
Time Frame: For each participant, the first occurrence of the outcome after randomization up until the efficacy cut-off date (08-Sep-2019) was considered. The mean survival time until ECOD was 1188.48 days
Population: Intention-to-treat analysis set (ITT Set): Comprised all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Rivaroxaban 2.5 mg Bid + Aspirin 100 mg od | Rivaroxaban Placebo Bid + Aspirin 100 mg od
Number analyzed (Participants) | 3286 | 3278
Participants | 321 | 297
Statistical Analysis 1: Comparison: Rivaroxaban 2.5 mg Bid + Aspirin 100 mg od vs Rivaroxaban Placebo Bid + Aspirin 100 mg od; Test type: Superiority; p = 0.8322, Log Rank — [p-value comment as in outcome 3, analysis 1]; Hazard Ratio (HR) = 1.08, 95% CI 2-sided [0.92 to 1.27]

9. Secondary Outcome: Number of Participants With Venous Thromboembolic (VTE) Events
Description: Venous thromboembolic events were reported by investigator only.
Time Frame: For each participant, the first occurrence of the outcome after randomization up until the efficacy cut-off date (08-Sep-2019) was considered. The mean survival time until ECOD was 1187.65 days
Population: Intention-to-treat analysis set (ITT Set): Comprised all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Rivaroxaban 2.5 mg Bid + Aspirin 100 mg od | Rivaroxaban Placebo Bid + Aspirin 100 mg od
Number analyzed (Participants) | 3286 | 3278
Participants | 25 | 41
Statistical Analysis 1: Comparison: Rivaroxaban 2.5 mg Bid + Aspirin 100 mg od vs Rivaroxaban Placebo Bid + Aspirin 100 mg od; Test type: Superiority; p = 0.0235, Log Rank — [p-value comment as in outcome 3, analysis 1]; Hazard Ratio (HR) = 0.61, 95% CI 2-sided [0.37 to 1.00]

10. Secondary Outcome: Secondary Safety Outcome: Number of Participants With ISTH (International Society on Thrombosis and Haemostasis) Major Bleeding
Description: Only the first occurrence of the outcome event under analysis within the data scope from a participant is considered.
Time Frame: For each participant, the first occurrence of the major bleeding events according to the ISTH classification after randomization up until 2 days after permanent stop of study drug (rivaroxaban or rivaroxaban placebo).
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Rivaroxaban 2.5 mg Bid + Aspirin 100 mg od | Rivaroxaban Placebo Bid + Aspirin 100 mg od
Number analyzed (Participants) | 3256 | 3248
Participants | 140 | 100
Statistical Analysis 1: Comparison: Rivaroxaban 2.5 mg Bid + Aspirin 100 mg od vs Rivaroxaban Placebo Bid + Aspirin 100 mg od; Test type: Other; p = 0.0068, Log Rank; Hazard Ratio (HR) = 1.42, 95% CI 2-sided [1.10 to 1.84]

11. Secondary Outcome: Secondary Safety Outcome: Number of Participants With BARC (Bleeding Academic Research Consortium) Type 3b and Above Bleeding Events
Description: Only the first occurrence of the outcome event under analysis within the data scope from a participant is considered
Time Frame: For each participant, the first occurrence of the type 3b and above bleeding events according to the BARC classification after randomization up until 2 days after permanent stop of study drug (rivaroxaban or rivaroxaban placebo)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Rivaroxaban 2.5 mg Bid + Aspirin 100 mg od | Rivaroxaban Placebo Bid + Aspirin 100 mg od
Number analyzed (Participants) | 3256 | 3248
Participants | 93 | 73
Statistical Analysis 1: Comparison: Rivaroxaban 2.5 mg Bid + Aspirin 100 mg od vs Rivaroxaban Placebo Bid + Aspirin 100 mg od; Test type: Other; p = 0.0979, Log Rank; Hazard Ratio (HR) = 1.29, 95% CI 2-sided [0.95 to 1.76]

ADVERSE EVENTS:
Time Frame: From randomization until 2 days following permanent discontinuation of the study drug
Arm/Group | Rivaroxaban 2.5 mg Bid + Aspirin 100 mg od | Rivaroxaban Placebo Bid + Aspirin 100 mg od
All-Cause Mortality (participants affected / at risk) | 327/3256 | 304/3248
Serious Adverse Events (participants affected / at risk) | 948/3256 | 927/3248
Other Adverse Events (participants affected / at risk) | 725/3256 | 729/3248
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rivaroxaban 2.5 mg Bid + Aspirin 100 mg od (N=3256) | Rivaroxaban Placebo Bid + Aspirin 100 mg od (N=3248)
Anaemia (Blood and lymphatic system disorders) | 14 (16) | 10 (13)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 4 (4) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Microcytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Normocytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Nephrogenic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Blood loss anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 10 (11) | 10 (10)
Angina unstable (Cardiac disorders) | 2 (2) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 2 (2) | 0 (0)
Arrhythmia (Cardiac disorders) | 3 (3) | 1 (1)
Arrhythmia supraventricular (Cardiac disorders) | 0 (0) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 2 (2) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 19 (19) | 20 (21)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 3 (3) | 2 (2)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 2 (2)
Bradycardia (Cardiac disorders) | 2 (2) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure (Cardiac disorders) | 14 (16) | 14 (15)
Cardiac failure acute (Cardiac disorders) | 3 (3) | 6 (6)
Cardiac failure chronic (Cardiac disorders) | 6 (8) | 3 (4)
Cardiac failure congestive (Cardiac disorders) | 10 (11) | 8 (8)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 2 (2) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 1 (1)
Coronary artery disease (Cardiac disorders) | 15 (18) | 21 (21)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 4 (4) | 2 (2)
Cyanosis (Cardiac disorders) | 1 (1) | 0 (0)
Hypertensive heart disease (Cardiac disorders) | 0 (0) | 2 (2)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 2 (2) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 2 (3)
Pericardial haemorrhage (Cardiac disorders) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Right ventricular failure (Cardiac disorders) | 0 (0) | 2 (2)
Sinus arrest (Cardiac disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 3 (3) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Ischaemic cardiomyopathy (Cardiac disorders) | 1 (3) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 1 (1)
Congestive cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Acute left ventricular failure (Cardiac disorders) | 2 (2) | 1 (1)
Supraventricular tachyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Stress cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 2 (2)
Congenital bladder neck obstruction (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Hydrocele (Congenital, familial and genetic disorders) | 1 (1) | 1 (1)
Phimosis (Congenital, familial and genetic disorders) | 0 (0) | 2 (2)
Adenomatous polyposis coli (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Deafness (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 2 (2)
Sudden hearing loss (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Goitre (Endocrine disorders) | 2 (2) | 1 (1)
Thyroid mass (Endocrine disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 8 (9) | 8 (10)
Cataract subcapsular (Eye disorders) | 1 (1) | 0 (0)
Diabetic retinopathy (Eye disorders) | 3 (3) | 2 (2)
Eyelid ptosis (Eye disorders) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 2 (2) | 0 (0)
Iridocyclitis (Eye disorders) | 0 (0) | 1 (1)
Macular degeneration (Eye disorders) | 1 (1) | 0 (0)
Macular oedema (Eye disorders) | 1 (1) | 0 (0)
Myopia (Eye disorders) | 0 (0) | 1 (1)
Retinal detachment (Eye disorders) | 0 (0) | 1 (1)
Retinal haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Vitreous haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Macular hole (Eye disorders) | 1 (1) | 0 (0)
Detachment of macular retinal pigment epithelium (Eye disorders) | 0 (0) | 1 (1)
Vitreoretinal traction syndrome (Eye disorders) | 1 (1) | 1 (1)
Macular detachment (Eye disorders) | 0 (0) | 1 (1)
Abdominal adhesions (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal mass (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (4) | 2 (2)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chronic gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Colitis ischaemic (Gastrointestinal disorders) | 2 (2) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dental alveolar anomaly (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diaphragmatic hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 3 (3) | 1 (1)
Gallstone ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric polyps (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 3 (3) | 1 (1)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 3 (3) | 1 (1)
Gastritis erosive (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal necrosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 2 (2) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 2 (2) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 4 (4) | 4 (4)
Intestinal angina (Gastrointestinal disorders) | 0 (0) | 1 (2)
Intestinal ischaemia (Gastrointestinal disorders) | 4 (4) | 3 (3)
Intestinal obstruction (Gastrointestinal disorders) | 3 (3) | 3 (3)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Intestinal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (3)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 4 (4) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 4 (5)
Pancreatitis chronic (Gastrointestinal disorders) | 0 (0) | 4 (4)
Pancreatitis necrotising (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peptic ulcer perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Periodontal disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 3 (3)
Small intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tooth loss (Gastrointestinal disorders) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 2 (2) | 1 (1)
Umbilical hernia, obstructive (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Volvulus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
Pancreatic mass (Gastrointestinal disorders) | 0 (0) | 1 (1)
Subileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0)
Mechanical ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric antral vascular ectasia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 10 (10) | 4 (4)
Oedematous pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Alcoholic pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (3)
Enterovesical fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatic duct stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal incarcerated hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Obstructive pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 4 (4) | 3 (3)
Crepitations (General disorders) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 1 (1)
Granuloma (General disorders) | 1 (1) | 0 (0)
Hernia (General disorders) | 0 (0) | 1 (1)
Impaired healing (General disorders) | 3 (3) | 7 (7)
Oedema (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 2 (2)
Pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 2 (3)
General physical health deterioration (General disorders) | 2 (2) | 1 (1)
Puncture site haemorrhage (General disorders) | 1 (1) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0)
Organ failure (General disorders) | 1 (1) | 0 (0)
Inflammation (General disorders) | 1 (1) | 1 (1)
Drug intolerance (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 3 (3) | 3 (3)
Vascular stent thrombosis (General disorders) | 0 (0) | 1 (1)
Stent-graft endoleak (General disorders) | 1 (1) | 0 (0)
Vascular stent occlusion (General disorders) | 1 (1) | 2 (2)
Vascular stent stenosis (General disorders) | 11 (11) | 8 (10)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 2 (2)
Vascular device occlusion (General disorders) | 0 (0) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 3 (4) | 2 (3)
Cholangitis (Hepatobiliary disorders) | 1 (2) | 3 (6)
Cholangitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 7 (7) | 3 (3)
Cholecystitis acute (Hepatobiliary disorders) | 2 (2) | 12 (12)
Cholelithiasis (Hepatobiliary disorders) | 2 (2) | 1 (1)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cirrhosis alcoholic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 3 (3) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 2 (2) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatorenal syndrome (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bile duct obstruction (Hepatobiliary disorders) | 0 (0) | 3 (3)
Biliary dyskinesia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Steatohepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Primary biliary cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 2 (2)
Hypersensitivity (Immune system disorders) | 1 (1) | 1 (1)
Abscess (Infections and infestations) | 1 (1) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 4 (4) | 5 (5)
Arteriosclerotic gangrene (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Blister infected (Infections and infestations) | 0 (0) | 1 (1)
Bronchiolitis (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 2 (2) | 1 (1)
Carbuncle (Infections and infestations) | 0 (0) | 1 (2)
Cellulitis (Infections and infestations) | 19 (19) | 18 (20)
Cellulitis gangrenous (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 2 (2) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Diabetic gangrene (Infections and infestations) | 2 (2) | 2 (2)
Diarrhoea infectious (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 4 (4) | 5 (5)
Ear infection (Infections and infestations) | 0 (0) | 1 (2)
Eczema infected (Infections and infestations) | 1 (1) | 0 (0)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0)
Epididymitis (Infections and infestations) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 1 (1) | 10 (11)
Escherichia sepsis (Infections and infestations) | 1 (1) | 0 (0)
Fournier's gangrene (Infections and infestations) | 0 (0) | 1 (1)
Fungal cystitis (Infections and infestations) | 0 (0) | 1 (1)
Fungal skin infection (Infections and infestations) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 16 (18) | 20 (22)
Gastroenteritis (Infections and infestations) | 3 (3) | 2 (2)
Gastroenteritis salmonella (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 2 (2) | 0 (0)
Infected skin ulcer (Infections and infestations) | 6 (6) | 4 (4)
Influenza (Infections and infestations) | 2 (2) | 0 (0)
Localised infection (Infections and infestations) | 19 (19) | 11 (11)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 2 (3)
Lymphangitis (Infections and infestations) | 1 (1) | 0 (0)
Mastoiditis (Infections and infestations) | 1 (1) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Ophthalmic herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Orchitis (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 11 (15) | 12 (14)
Osteomyelitis chronic (Infections and infestations) | 3 (3) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 1 (1)
Perinephric abscess (Infections and infestations) | 1 (2) | 0 (0)
Periodontitis (Infections and infestations) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 1 (1) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 40 (49) | 45 (50)
Postoperative wound infection (Infections and infestations) | 27 (28) | 25 (26)
Pseudomembranous colitis (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 2 (2) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 3 (3)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 12 (12) | 13 (13)
Septic shock (Infections and infestations) | 1 (1) | 5 (5)
Sinusitis (Infections and infestations) | 0 (0) | 2 (2)
Skin infection (Infections and infestations) | 2 (2) | 2 (2)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 13 (17) | 11 (13)
Wound infection (Infections and infestations) | 17 (19) | 15 (16)
Urosepsis (Infections and infestations) | 0 (0) | 5 (5)
Streptococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Scrotal abscess (Infections and infestations) | 1 (1) | 1 (1)
Groin abscess (Infections and infestations) | 3 (3) | 0 (0)
Abscess limb (Infections and infestations) | 6 (8) | 5 (5)
Groin infection (Infections and infestations) | 1 (1) | 1 (1)
Lymph gland infection (Infections and infestations) | 1 (1) | 0 (0)
Periumbilical abscess (Infections and infestations) | 0 (0) | 1 (1)
Burn infection (Infections and infestations) | 1 (2) | 0 (0)
Haematoma infection (Infections and infestations) | 1 (1) | 1 (1)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 2 (2)
Perineal abscess (Infections and infestations) | 2 (2) | 0 (0)
Arthritis bacterial (Infections and infestations) | 2 (2) | 2 (2)
Abdominal infection (Infections and infestations) | 1 (1) | 0 (0)
Graft infection (Infections and infestations) | 1 (1) | 0 (0)
Gastric infection (Infections and infestations) | 0 (0) | 1 (1)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 3 (4) | 2 (2)
Infected lymphocele (Infections and infestations) | 2 (2) | 0 (0)
Intervertebral discitis (Infections and infestations) | 1 (1) | 1 (1)
Diabetic foot infection (Infections and infestations) | 1 (3) | 6 (6)
Pneumonia bacterial (Infections and infestations) | 2 (2) | 3 (3)
Arthritis infective (Infections and infestations) | 1 (1) | 0 (0)
Extradural abscess (Infections and infestations) | 1 (1) | 0 (0)
Soft tissue infection (Infections and infestations) | 2 (2) | 3 (3)
Respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Cholecystitis infective (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 2 (2) | 2 (2)
Cystitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Dermo-hypodermitis (Infections and infestations) | 1 (1) | 0 (0)
Post procedural sepsis (Infections and infestations) | 0 (0) | 1 (1)
Superinfection bacterial (Infections and infestations) | 0 (0) | 1 (1)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0)
Bone abscess (Infections and infestations) | 1 (1) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 0 (0) | 1 (1)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Infected seroma (Infections and infestations) | 1 (1) | 0 (0)
Medical device site infection (Infections and infestations) | 1 (2) | 0 (0)
Medical device site joint infection (Infections and infestations) | 0 (0) | 3 (4)
Perineal cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Vascular device infection (Infections and infestations) | 2 (3) | 2 (2)
Complicated appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Large intestine infection (Infections and infestations) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 2 (2) | 3 (4)
Brain herniation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Failure to anastomose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 5 (5) | 2 (2)
Femoral neck fracture (Injury, poisoning and procedural complications) | 4 (4) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 10 (10) | 12 (12)
Fibula fracture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fractured sacrum (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 5 (5) | 5 (5)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Intentional overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Open fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Penetrating abdominal trauma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Rib fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 1 (1) | 1 (2)
Skull fractured base (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 4 (5)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Traumatic ulcer (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 4 (4) | 3 (3)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Vascular graft occlusion (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Traumatic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 2 (2) | 4 (4)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Anastomotic stenosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Graft thrombosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound necrosis (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Coronary artery restenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post laminectomy syndrome (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Underdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular procedure complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural bile leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural discharge (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Chemical burn of skin (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 2 (3) | 4 (4)
Chest injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Post procedural oedema (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Vascular graft complication (Injury, poisoning and procedural complications) | 5 (5) | 1 (1)
Cerebral hyperperfusion syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Bone contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Periprosthetic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Peripheral arterial reocclusion (Injury, poisoning and procedural complications) | 4 (6) | 2 (3)
Spinal column injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pubis fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Peripheral artery restenosis (Injury, poisoning and procedural complications) | 16 (22) | 15 (18)
Meniscus injury (Injury, poisoning and procedural complications) | 2 (2) | 4 (4)
Skin scar contracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural intestinal perforation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular graft stenosis (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Vascular graft restenosis (Injury, poisoning and procedural complications) | 0 (0) | 2 (4)
Vascular access site haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arterial bypass thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arterial bypass occlusion (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Arterial bypass stenosis (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Foreign body in gastrointestinal tract (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 0 (0) | 1 (1)
Blood potassium increased (Investigations) | 1 (1) | 1 (1)
Blood pressure increased (Investigations) | 0 (0) | 1 (1)
Cardiovascular function test abnormal (Investigations) | 0 (0) | 1 (2)
Cystoscopy (Investigations) | 1 (1) | 0 (0)
Immunoglobulins decreased (Investigations) | 1 (1) | 0 (0)
Carbohydrate antigen 19-9 increased (Investigations) | 1 (1) | 0 (0)
Cardiac stress test abnormal (Investigations) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0)
Vascular test (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 6 (6) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 6 (6) | 8 (9)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (4)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 3 (3) | 6 (7)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (3) | 5 (8)
Ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic disorder (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypophagia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 3 (3) | 5 (6)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Bone disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Bone formation increased (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Fracture nonunion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Jaw cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (4)
Metatarsalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Osteitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 14 (18) | 13 (14)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (6) | 14 (15)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (3) | 4 (4)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 6 (7) | 6 (7)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Spondyloarthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Vertebral column mass (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acquired claw toe (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Ligament disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Soft tissue disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Bone loss (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3)
Systemic scleroderma (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 6 (6) | 2 (2)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 7 (7)
Benign laryngeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 4 (4)
Bladder cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Bone cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Central nervous system lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Chronic myelomonocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 4 (4)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Follicular thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 4 (4)
Gastric cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastric cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 3 (3)
Laryngeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 3 (3)
Lung adenocarcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung adenocarcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Lung carcinoma cell type unspecified recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Lung squamous cell carcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Metastases to neck (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 1 (1)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
Oesophageal carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Oropharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
Papillary serous endometrial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pleural mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Rectal cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Rectal cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Small cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
Rectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 3 (3)
Salivary gland adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oesophageal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 1 (1)
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (8) | 14 (16)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic carcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 (9) | 2 (2)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Thymoma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Respiratory tract neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Adrenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hodgkin's disease stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 1 (1)
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 4 (4)
Rectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gingival cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (3) | 0 (0)
Head and neck cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Inflammatory pseudotumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenolymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung squamous cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ductal adenocarcinoma of pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant genitourinary tract neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant neoplasm papilla of Vater (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastrointestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Skin squamous cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 22 (23) | 24 (26)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1) | 2 (2)
Cerebral atrophy (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Dementia (Nervous system disorders) | 3 (3) | 2 (2)
Diabetic neuropathy (Nervous system disorders) | 2 (2) | 2 (2)
Dizziness (Nervous system disorders) | 5 (5) | 3 (3)
Dizziness postural (Nervous system disorders) | 1 (1) | 0 (0)
Drop attacks (Nervous system disorders) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1) | 1 (1)
Guillain-Barre syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Hemiparesis (Nervous system disorders) | 0 (0) | 1 (1)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1)
Intracranial aneurysm (Nervous system disorders) | 0 (0) | 1 (1)
Mental impairment (Nervous system disorders) | 1 (1) | 0 (0)
Myelopathy (Nervous system disorders) | 1 (1) | 2 (3)
Nerve compression (Nervous system disorders) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 2 (2)
Parkinsonism (Nervous system disorders) | 0 (0) | 1 (1)
Polyneuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 2 (2) | 1 (1)
Sciatica (Nervous system disorders) | 2 (2) | 4 (4)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Spinal claudication (Nervous system disorders) | 1 (1) | 1 (1)
Status epilepticus (Nervous system disorders) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 9 (9) | 11 (12)
Tension headache (Nervous system disorders) | 1 (1) | 0 (0)
Tonic convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Vertebral artery stenosis (Nervous system disorders) | 0 (0) | 1 (1)
Carotid artery occlusion (Nervous system disorders) | 0 (0) | 1 (1)
Cervical radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Lumbar radiculopathy (Nervous system disorders) | 1 (2) | 0 (0)
Facial paresis (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Restless legs syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Putamen haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Cranial nerve disorder (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Parkinson's disease (Nervous system disorders) | 1 (1) | 1 (1)
Carotid artery disease (Nervous system disorders) | 1 (1) | 1 (1)
Vascular encephalopathy (Nervous system disorders) | 1 (1) | 1 (1)
Pseudoradicular syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Brain injury (Nervous system disorders) | 1 (1) | 0 (0)
Colloid brain cyst (Nervous system disorders) | 0 (0) | 1 (1)
Sacral radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Acute psychosis (Psychiatric disorders) | 0 (0) | 1 (1)
Alcohol abuse (Psychiatric disorders) | 1 (1) | 1 (1)
Alcoholism (Psychiatric disorders) | 1 (2) | 0 (0)
Completed suicide (Psychiatric disorders) | 4 (4) | 0 (0)
Depression (Psychiatric disorders) | 3 (3) | 5 (5)
Drug abuse (Psychiatric disorders) | 0 (0) | 1 (1)
Intentional self-injury (Psychiatric disorders) | 1 (1) | 0 (0)
Organic brain syndrome (Psychiatric disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1) | 4 (4)
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 (0) | 1 (1)
Transient psychosis (Psychiatric disorders) | 1 (1) | 0 (0)
Calculus bladder (Renal and urinary disorders) | 3 (3) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 2 (2)
Pelvi-ureteric obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal artery stenosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 4 (4) | 0 (0)
Renal failure (Renal and urinary disorders) | 6 (8) | 3 (3)
Ureteric fistula (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 2 (2)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 3 (3) | 3 (3)
Chronic kidney disease (Renal and urinary disorders) | 5 (5) | 2 (2)
Urethral stenosis (Renal and urinary disorders) | 1 (1) | 2 (3)
Acute kidney injury (Renal and urinary disorders) | 9 (9) | 17 (17)
End stage renal disease (Renal and urinary disorders) | 1 (1) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 3 (3) | 2 (2)
Cervical polyp (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pelvic prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Spermatocele (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterine prolapse (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Vulvar dysplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Prostatic obstruction (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vulval eczema (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 16 (23) | 9 (12)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 6 (6)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 6 (6)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 2 (2)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (4)
Sinus polyp (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pharyngeal lesion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tonsillar cyst (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic respiratory disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute interstitial pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pemphigoid (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Pemphigus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Skin ulcer (Skin and subcutaneous tissue disorders) | 10 (11) | 12 (14)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Diabetic foot (Skin and subcutaneous tissue disorders) | 9 (9) | 9 (11)
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Ischaemic skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Myxoid cyst (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Disease risk factor (Social circumstances) | 0 (0) | 1 (1)
Bladder calculus removal (Surgical and medical procedures) | 0 (0) | 1 (1)
Blepharoplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Carotid endarterectomy (Surgical and medical procedures) | 1 (1) | 1 (1)
Foot amputation (Surgical and medical procedures) | 1 (1) | 0 (0)
Knee arthroplasty (Surgical and medical procedures) | 0 (0) | 2 (2)
Umbilical hernia repair (Surgical and medical procedures) | 1 (1) | 0 (0)
Vitrectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Radical prostatectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Diabetes mellitus management (Surgical and medical procedures) | 0 (0) | 1 (1)
Transurethral bladder resection (Surgical and medical procedures) | 0 (0) | 1 (1)
Peripheral revascularisation (Surgical and medical procedures) | 0 (0) | 1 (1)
Brain tumour operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Cystoprostatectomy (Surgical and medical procedures) | 1 (1) | 1 (1)
Peripheral artery angioplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Amputation (Surgical and medical procedures) | 1 (1) | 0 (0)
Bladder polypectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Bladder neoplasm surgery (Surgical and medical procedures) | 1 (1) | 1 (1)
Limb reconstructive surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Peripheral artery bypass (Surgical and medical procedures) | 0 (0) | 1 (1)
Peripheral artery stent insertion (Surgical and medical procedures) | 1 (1) | 0 (0)
Eventration repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Aortic aneurysm (Vascular disorders) | 2 (3) | 4 (4)
Aortic dissection (Vascular disorders) | 1 (1) | 0 (0)
Aortic stenosis (Vascular disorders) | 6 (6) | 3 (3)
Arteriovenous fistula (Vascular disorders) | 0 (0) | 1 (1)
Circulatory collapse (Vascular disorders) | 1 (1) | 2 (2)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 5 (5)
Hypertensive crisis (Vascular disorders) | 5 (5) | 6 (8)
Hypotension (Vascular disorders) | 4 (4) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 0 (0)
Intermittent claudication (Vascular disorders) | 43 (51) | 52 (58)
Lymphoedema (Vascular disorders) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)
Peripheral coldness (Vascular disorders) | 0 (0) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 34 (44) | 29 (46)
Peripheral vascular disorder (Vascular disorders) | 3 (4) | 5 (5)
Poor peripheral circulation (Vascular disorders) | 1 (1) | 1 (1)
Renovascular hypertension (Vascular disorders) | 1 (1) | 0 (0)
Temporal arteritis (Vascular disorders) | 1 (1) | 0 (0)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 1 (1)
Varicose vein (Vascular disorders) | 1 (1) | 2 (2)
Lymphocele (Vascular disorders) | 1 (1) | 2 (2)
Dry gangrene (Vascular disorders) | 2 (3) | 3 (3)
Subclavian artery stenosis (Vascular disorders) | 0 (0) | 1 (1)
Lymphorrhoea (Vascular disorders) | 2 (2) | 0 (0)
Iliac artery stenosis (Vascular disorders) | 4 (4) | 3 (3)
Vascular stenosis (Vascular disorders) | 0 (0) | 1 (1)
Peripheral artery aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Peripheral artery occlusion (Vascular disorders) | 7 (9) | 9 (10)
Hypertensive emergency (Vascular disorders) | 1 (1) | 0 (0)
Hypertensive urgency (Vascular disorders) | 0 (0) | 1 (1)
Venous occlusion (Vascular disorders) | 1 (1) | 0 (0)
Angiopathy (Vascular disorders) | 1 (1) | 0 (0)
Extremity necrosis (Vascular disorders) | 12 (14) | 8 (9)
Peripheral embolism (Vascular disorders) | 1 (1) | 2 (2)
Peripheral arterial occlusive disease (Vascular disorders) | 125 (156) | 130 (182)
Arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1)
Ischaemic limb pain (Vascular disorders) | 0 (0) | 1 (1)
Lymphatic fistula (Vascular disorders) | 0 (0) | 3 (3)
Peripheral artery stenosis (Vascular disorders) | 25 (29) | 14 (17)
Peripheral artery thrombosis (Vascular disorders) | 2 (2) | 2 (2)
Peripheral venous disease (Vascular disorders) | 1 (1) | 0 (0)
Device breakage (Product Issues) | 2 (2) | 0 (0)
Device dislocation (Product Issues) | 1 (1) | 0 (0)
Device occlusion (Product Issues) | 0 (0) | 1 (1)
Patient-device incompatibility (Product Issues) | 1 (1) | 0 (0)
Device battery issue (Product Issues) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rivaroxaban 2.5 mg Bid + Aspirin 100 mg od (N=3256) | Rivaroxaban Placebo Bid + Aspirin 100 mg od (N=3248)
Anaemia (Blood and lymphatic system disorders) | 29 (29) | 23 (23)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 8 (9) | 3 (3)
Angina pectoris (Cardiac disorders) | 9 (10) | 7 (7)
Atrial fibrillation (Cardiac disorders) | 31 (33) | 48 (49)
Atrial flutter (Cardiac disorders) | 7 (7) | 2 (2)
Cardiac failure (Cardiac disorders) | 3 (4) | 7 (7)
Coronary artery disease (Cardiac disorders) | 12 (13) | 9 (9)
Myocardial ischaemia (Cardiac disorders) | 6 (6) | 1 (1)
Palpitations (Cardiac disorders) | 3 (3) | 4 (4)
Sinus tachycardia (Cardiac disorders) | 4 (4) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 4 (5) | 3 (3)
Vertigo (Ear and labyrinth disorders) | 7 (7) | 11 (13)
Cataract (Eye disorders) | 14 (17) | 9 (9)
Diabetic retinopathy (Eye disorders) | 4 (4) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 6 (7) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 6 (6) | 6 (6)
Abdominal pain upper (Gastrointestinal disorders) | 19 (19) | 15 (16)
Constipation (Gastrointestinal disorders) | 11 (11) | 13 (13)
Diarrhoea (Gastrointestinal disorders) | 23 (24) | 22 (22)
Diverticulum intestinal (Gastrointestinal disorders) | 1 (1) | 4 (4)
Duodenal ulcer (Gastrointestinal disorders) | 4 (4) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 15 (16) | 8 (8)
Gastric ulcer (Gastrointestinal disorders) | 4 (4) | 5 (5)
Gastritis (Gastrointestinal disorders) | 15 (15) | 8 (8)
Gastritis erosive (Gastrointestinal disorders) | 2 (2) | 5 (5)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 8 (8) | 8 (9)
Hiatus hernia (Gastrointestinal disorders) | 4 (4) | 2 (2)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 5 (5)
Nausea (Gastrointestinal disorders) | 14 (14) | 10 (10)
Vomiting (Gastrointestinal disorders) | 7 (7) | 13 (13)
Large intestine polyp (Gastrointestinal disorders) | 6 (6) | 4 (4)
Asthenia (General disorders) | 6 (6) | 4 (4)
Chest discomfort (General disorders) | 6 (6) | 1 (1)
Chest pain (General disorders) | 11 (12) | 16 (16)
Fatigue (General disorders) | 11 (11) | 12 (14)
Gait disturbance (General disorders) | 5 (5) | 2 (2)
Impaired healing (General disorders) | 4 (4) | 2 (2)
Oedema peripheral (General disorders) | 16 (17) | 20 (21)
Peripheral swelling (General disorders) | 9 (10) | 10 (10)
Non-cardiac chest pain (General disorders) | 5 (5) | 3 (3)
Vascular stent stenosis (General disorders) | 9 (10) | 10 (10)
Hepatic steatosis (Hepatobiliary disorders) | 4 (4) | 2 (2)
Hypersensitivity (Immune system disorders) | 1 (1) | 5 (5)
Bronchitis (Infections and infestations) | 15 (17) | 17 (21)
Cellulitis (Infections and infestations) | 10 (11) | 6 (7)
Gangrene (Infections and infestations) | 5 (5) | 2 (2)
Herpes zoster (Infections and infestations) | 5 (5) | 7 (7)
Influenza (Infections and infestations) | 10 (11) | 7 (8)
Localised infection (Infections and infestations) | 11 (11) | 7 (7)
Nasopharyngitis (Infections and infestations) | 21 (23) | 30 (32)
Osteomyelitis (Infections and infestations) | 4 (4) | 1 (1)
Pneumonia (Infections and infestations) | 9 (9) | 14 (14)
Postoperative wound infection (Infections and infestations) | 9 (9) | 9 (9)
Sinusitis (Infections and infestations) | 6 (6) | 3 (4)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 2 (2)
Urinary tract infection (Infections and infestations) | 22 (23) | 21 (27)
Wound infection (Infections and infestations) | 9 (9) | 4 (4)
Respiratory tract infection viral (Infections and infestations) | 2 (2) | 4 (4)
Respiratory tract infection (Infections and infestations) | 5 (5) | 2 (3)
Fall (Injury, poisoning and procedural complications) | 6 (6) | 6 (6)
Foot fracture (Injury, poisoning and procedural complications) | 5 (5) | 2 (2)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 5 (5)
Rib fracture (Injury, poisoning and procedural complications) | 2 (2) | 6 (6)
Muscle strain (Injury, poisoning and procedural complications) | 4 (4) | 3 (3)
Contusion (Injury, poisoning and procedural complications) | 9 (11) | 10 (11)
Limb injury (Injury, poisoning and procedural complications) | 11 (11) | 11 (11)
Peripheral artery restenosis (Injury, poisoning and procedural complications) | 5 (8) | 6 (8)
Meniscus injury (Injury, poisoning and procedural complications) | 2 (2) | 4 (4)
Arterial bypass occlusion (Injury, poisoning and procedural complications) | 2 (2) | 5 (5)
Blood pressure increased (Investigations) | 4 (5) | 6 (6)
Haemoglobin decreased (Investigations) | 5 (5) | 2 (2)
Diabetes mellitus (Metabolism and nutrition disorders) | 6 (6) | 12 (12)
Gout (Metabolism and nutrition disorders) | 5 (5) | 11 (11)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 4 (4)
Vitamin D deficiency (Metabolism and nutrition disorders) | 5 (5) | 1 (1)
Dyslipidaemia (Metabolism and nutrition disorders) | 1 (1) | 5 (5)
Decreased appetite (Metabolism and nutrition disorders) | 6 (6) | 4 (4)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 13 (13) | 7 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 18 (19) | 32 (37)
Back pain (Musculoskeletal and connective tissue disorders) | 23 (25) | 30 (33)
Bursitis (Musculoskeletal and connective tissue disorders) | 5 (6) | 7 (7)
Joint swelling (Musculoskeletal and connective tissue disorders) | 6 (6) | 2 (2)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 5 (6) | 2 (4)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 13 (14) | 13 (16)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 (4) | 5 (6)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 10 (10) | 11 (11)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (6) | 4 (4)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 12 (12) | 14 (14)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 47 (58) | 52 (53)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (3)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (6)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 7 (7) | 5 (5)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 4 (4) | 5 (5)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 4 (4)
Carotid artery stenosis (Nervous system disorders) | 3 (3) | 8 (10)
Carpal tunnel syndrome (Nervous system disorders) | 2 (2) | 6 (6)
Diabetic neuropathy (Nervous system disorders) | 3 (3) | 4 (4)
Dizziness (Nervous system disorders) | 23 (27) | 26 (28)
Headache (Nervous system disorders) | 18 (20) | 19 (21)
Hypoaesthesia (Nervous system disorders) | 6 (7) | 8 (9)
Neuropathy peripheral (Nervous system disorders) | 5 (5) | 1 (1)
Paraesthesia (Nervous system disorders) | 4 (4) | 9 (9)
Sciatica (Nervous system disorders) | 6 (6) | 13 (14)
Syncope (Nervous system disorders) | 3 (3) | 9 (10)
Delirium (Psychiatric disorders) | 0 (0) | 4 (4)
Depression (Psychiatric disorders) | 11 (12) | 14 (14)
Dysuria (Renal and urinary disorders) | 3 (3) | 4 (4)
Haematuria (Renal and urinary disorders) | 4 (4) | 2 (2)
Renal failure (Renal and urinary disorders) | 2 (2) | 5 (6)
Renal impairment (Renal and urinary disorders) | 4 (5) | 6 (6)
Chronic kidney disease (Renal and urinary disorders) | 8 (8) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 7 (8) | 4 (4)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 5 (5) | 9 (9)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 4 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 14 (14)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 15 (15)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9 (14) | 3 (3)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4)
Ecchymosis (Skin and subcutaneous tissue disorders) | 5 (5) | 2 (2)
Eczema (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (4)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 5 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 10 (11) | 7 (7)
Rash (Skin and subcutaneous tissue disorders) | 16 (16) | 18 (20)
Skin ulcer (Skin and subcutaneous tissue disorders) | 16 (17) | 18 (18)
Urticaria (Skin and subcutaneous tissue disorders) | 7 (7) | 5 (5)
Diabetic foot (Skin and subcutaneous tissue disorders) | 6 (6) | 1 (1)
Tooth extraction (Surgical and medical procedures) | 6 (7) | 5 (5)
Cataract operation (Surgical and medical procedures) | 5 (6) | 8 (10)
Hypertension (Vascular disorders) | 49 (54) | 50 (56)
Hypertensive crisis (Vascular disorders) | 11 (13) | 13 (15)
Hypotension (Vascular disorders) | 7 (7) | 3 (3)
Intermittent claudication (Vascular disorders) | 39 (48) | 43 (48)
Peripheral ischaemia (Vascular disorders) | 3 (3) | 11 (14)
Peripheral vascular disorder (Vascular disorders) | 6 (8) | 5 (5)
Dry gangrene (Vascular disorders) | 1 (1) | 4 (4)
Peripheral artery occlusion (Vascular disorders) | 6 (6) | 12 (13)
Extremity necrosis (Vascular disorders) | 6 (7) | 5 (5)
Peripheral arterial occlusive disease (Vascular disorders) | 34 (45) | 31 (37)
Peripheral artery stenosis (Vascular disorders) | 13 (16) | 10 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-07-24): https://cdn.clinicaltrials.gov/large-docs/16/NCT02504216/SAP_000.pdf
  • Study Protocol (2017-03-21): https://cdn.clinicaltrials.gov/large-docs/16/NCT02504216/Prot_001.pdf